CLINICAL TRIAL: NCT06890234
Title: Clinical Applicability of Tissue Microdialysis for Early Assessment of Liver Graft Metabolism in Patients After Orthotopic Liver Transplantation
Brief Title: Tissue Microdialysis Monitoring of Liver Grafts
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Sergej Godec, Medical Doctor, intensive care specialist, University Medical Centre Ljubljana
Other Study IDs: 0120-505/2023/3; TP20230129 (Other Grant/Funding Number: UMC Ljubljana); TP20240197 (Other Grant/Funding Number: UMC Ljubljana)
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Liver Transplantation; Liver Graft Dysfunction; Tissue Metabolism
Keywords: microdialysis; liver graft monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples With DNA — Interstitial molecules in liver tissue with a molecular weight below 100 kDa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients (≥18 years old) who have undergone orthotopic liver transplantation

SUMMARY:
This study will investigate the dynamics of metabolic molecules sampled from human liver grafts during the early postoperative period using tissue microdialysis. The obtained tissue samples will be compared with standard liver function tests and dynamic functional liver assessment tests. The primary objective is to evaluate the clinical feasibility, utility, and non-inferiority of tissue microdialysis in comparison to current standard methods for monitoring liver grafts.

ELIGIBILITY:
Inclusion criteria:

* Adult patients aged between 18 and 65 years.
* Liver transplant candidates on the Slovenian liver transplant waiting list, matched with an available liver graft through the Eurotransplant system, and scheduled for the surgical procedure.
* Signed informed consent to participate in the microdialysis sampling research project, including consent to share the obtained samples with other research studies

Exclusion criteria:

* Patients under 18 or over 65 years of age.
* Refusal to participate in the study.
* Verbal withdrawal of consent at any point during the study, even if informed consent has been previously signed.
* Surgical contraindications preventing the insertion of a microdialysis catheter into the liver graft during the procedure.
* Surgical revision within 48 hours post-transplantation resulting in liver graft loss and removal.
* History of allergic reactions to radiographic contrast media.
* Death during the liver transplant procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant candidates satisfying the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The agreement between microdialysis-derived metabolite levels and conventional liver function tests | From the end of liver transplant surgery up to 5 days post-transplant
  The correlation between tissue microdialysis metabolites (glucose, pyruvate, lactate, glycerol, urea) and standard static and dynamic liver function tests (ALT, AST, bilirubin, INR, plasma lactate, plasma pyruvate, and indocyanine green [ICG] clearance) in the early post-transplant period.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Raw data, with only IPD used in the results publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and ending 3 years after the publication of results
Access Criteria: A proposal describing the planned analyses must be submitted, and a data sharing agreement must be signed. Documents should be submitted via email to sergej.godec@kclj.si.